CLINICAL TRIAL: NCT04290975
Title: Bridging the Childhood Epilepsy Treatment Gap in Africa (BRIDGE)
Brief Title: Bridging the Childhood Epilepsy Treatment Gap in Africa
Acronym: BRIDGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Aminu Kano Teaching Hospital (Other); Ahmadu Bello University Teaching Hospital (Other); Federal Neuro-Psychiatric Hospital, Kaduna (Unknown)
Responsible Party: Principal Investigator, Edwin Trevathan, Professor of Neurology and Pediatrics, Director of Vanderbilt Institute for Global Health, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 191283; PACTR202003864779691 (Registry Identifier: Pan African Clinical Trials Registry)
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Pediatric; Neurology; Nigeria; Task-shifting; Africa
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The basic framework of these studies is a cRCTin which 60 PHCs (clusters) will be randomly selected from about 399 eligible PHCs in three major cities in the Hausa-speaking areas of northern Nigeria -30 of about 167 PHCs in Kano, 15 of about 124 PHCs in Kaduna, and 15 of about 108 PHCs in Zaria. Half of the overall PHCs will be randomly assigned to the task-shifted care arm of the cRCT, in which epilepsy treatment and follow-up care is provided by a CHW. The other half will be assigned to "enhanced usual care" in which the care is provided by a physician and a CHW serves to record events and collect other standardized data.
Who Masked: Outcomes Assessor
Masking Description: Blinded physicians will evaluate outcomes for both arms of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-shifted arm (Experimental): In the task-shifted arm, all children will be prescribed anti-epileptic medication and receive follow-up care from a CHW, with a physician consult available to the CHW as needed.
  Interventions: Other: Task-shifting of follow-up care for pediatric epilepsy
- Enhanced usual care arm (Active Comparator): In the enhanced usual care arm, all children will be prescribed anti-epileptic medication and receive follow-up care from a physician, with a CHW collecting standardized data to mirror that of the intervention arm.
  Interventions: Other: Enhanced usual care for pediatric epilepsy

INTERVENTIONS:
Other: Task-shifting of follow-up care for pediatric epilepsy — For the intervention arm, follow-up care of children with epilepsy will be shifted to be performed primarily by Community Health Workers (CHWs) with specialized epilepsy training
  Arms: Task-shifted arm
Other: Enhanced usual care for pediatric epilepsy — For the intervention arm, follow-up care of children with epilepsy will be performed primarily by physicians, with CHWs serving to collect standardized data regarding outcomes
  Arms: Enhanced usual care arm

SUMMARY:
About half of the world's children with epilepsy do not receive treatment - known as the epilepsy treatment gap - with significantly higher rates (67%-90%) in low- and middle-income countries (LMICs). We will conduct the first cluster-randomized clinical trial (cRCT) to determine the efficacy, implementation, and cost-effectiveness of a novel intervention shifting childhood epilepsy care to epilepsy-trained community health extension workers in an effort to close the epilepsy treatment gap. This research will provide information to help extend epilepsy treatment to children in LMICs and worldwide who suffer from untreated seizures.

DETAILED DESCRIPTION:
Epilepsy is the most common severe neurological disorder among children. Most children with epilepsy, if treated, can live normal lives. Yet among the world's children living with epilepsy, about 80% of whom reside in low- and middle-income countries (LMICs), about half do not receive treatment; this is described as "the childhood epilepsy treatment gap." Among the LMICs of Africa, the childhood epilepsy treatment gap is about 67%-90% - unchanged for over twenty years. Although the World Health Organization (WHO) and other health agencies recommend that the epilepsy treatment gap be bridged by task shifting epilepsy care to community health extension workers (CHWs) in primary care settings, this recommendation has not been implemented on a large scale. This failure to scale up task shifting in epilepsy care is due to (a) inadequate evidence of efficacy of task-shifted epilepsy care, (b) a lack of methods and tools for implementing epilepsy task shifting, (c) inadequate understanding of task-shifted epilepsy care barriers, and (d) a lack of cost-effectiveness data for health policymakers. CHWs providing task-shifted epilepsy care must identify children with epilepsy, disadvantaged by stigma and unknown to the healthcare system, who are without access to neurologists or electroencephalograms (EEGs). An epilepsy screening tool in the local language (e.g., Hausa) is therefore essential for epilepsy diagnosis, seizure type classification, and medical management. Hausa, the most commonly spoken language in west Africa, with over 120 million Hausa speakers, is used in daily life, commerce, and education; our proposed study will be conducted in three major cities in Hausa-speaking Africa.

Funded by an R21 grant (R21TW010899) in preparation for this cluster-randomized clinical trial (cRCT), we developed and piloted in Kano, Nigeria (a) a scalable epilepsy training program for CHWs, (b) an epilepsy community education program in Hausa to facilitate screening, diagnosis and treatment; and (c) an epilepsy data management system. We also (d) validated an epilepsy screening, diagnosis, and seizure classification tool in Hausa, (e) demonstrated feasibility of screening and enrolling children in a cRCT of task-shifted epilepsy care, and (f) piloted a task-shifted epilepsy diagnosis and management protocol. We will now conduct the first cRCT of task-shifted childhood epilepsy care in Africa with the following specific aims:

1. Conduct a non-inferiority cRCT of a task-shifted childhood epilepsy care protocol compared to enhanced usual care (EUC) in three Hausa-speaking cities in northern Nigeria. We will enroll a maximum of 1800 children (age 6 mo, <18 yrs) with epilepsy across 60 randomly selected primary healthcare centers (PHCs) in Kano (30 PHCs), Kaduna (16 PHCs) and Zaria (14 PHCs). PHCs will be randomly assigned to intervention (task-shifted to CHWS childhood epilepsy care; 30 PHCs) or EUC (referral to a physician for epilepsy management; 30 PHCs). Primary outcome: we hypothesize that the proportion of children seizure-free for ≥ 6 months at 24 months follow-up (primary outcome) will be similar in the intervention and EUC arms. Secondary outcomes at 24 months include (a) percent seizure reduction from baseline, (b) time to next seizure after 3 months seizure-free, and (c) accuracy of epilepsy diagnosis and seizure type classification by CHWs compared to assessments by physician epilepsy specialists, blinded to the randomization arm.
2. Assess socio-behavioral and implementation outcomes among providers, parents/guardians and patients in the cRCT. Outcome measures include: (1) Difference in baseline, 12- and 24-month intervention acceptability, appropriateness, and feasibility measures among providers in the task-shifted intervention arm of the cRCT; (2) Difference in baseline, 12- and 24-month quality of life, epilepsy knowledge and stigma, and trust in the healthcare system and providers among participants; (3) Comparison of 12- and 24-month quality of life, knowledge and stigma and trust measures among participants in the intervention and control arms.
3. Determine the cost-effectiveness of the task-shifted epilepsy care intervention. Direct costs of the intervention and EUC will include personnel costs (including CHW epilepsy training) and expenses for diagnostic (EEG, brain imaging) and laboratory tests and anti-epileptic drugs. Indirect costs will include travel time and time away from work for parents/guardians and change in school attendance for patients. Cost-effectiveness will be expressed as US dollars per disability adjusted life year (DALY) averted.

This project will also establish a brain disorders clinical research network for Hausa-speaking Africa and provide data for health system leaders and policymakers to scale-up task-shifted childhood epilepsy care.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Kano or Kaduna states and living in the Kano, Zaria, or Kaduna metropolitan areas of northern Nigeria
* Parent or guardian provided informed consent for the screening questionnaire given to the parent/guardian
* Parent or guardian informed consent, plus assent for children >7 years able to provide assent, for epilepsy diagnostic evaluation if the screening for possible epilepsy is positive
* Diagnosed with possible epilepsy through initial screening, and then diagnosed with epilepsy upon further evaluation by an epilepsy-trained CHW working with the BRIDGE project, who may consult a BRIDGE physician for diagnostic questions
* Parent or guardian provided consent, and assent for children >7 years able to provide assent, for enrollment in the cRCT of task-shifted epilepsy care versus enhanced physician epilepsy care

Exclusion Criteria:

* Children who have previously been diagnosed with epilepsy and are currently enrolled in other care and treatment, or who have been treated for epilepsy within three months prior to screening
* Children who are currently receiving care by a neurologist or neurosurgeon for a serious brain disorder (e.g., brain tumor, stroke)
* Lack of informed consent, and/or lack of assent from children >7 years who are able to provide assent.Inability of the parent or guardian to communicate with healthcare providers in either Hausa or English
* Any child who screens positive for epilepsy, has epilepsy upon clinical evaluation, but does not live in Kano, Zaria, and Kaduna, and who is in the judgement of the parents and/or BRIDGE staff to be unable to comply with the study visits because of travel distance from home.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage seizure-free | Must be seizure-free for 6 or more months at the 24-month visit follow-up visit
  Percentage of children in each arm of the study who are seizure-free

SECONDARY OUTCOMES:
Reduction in seizure frequency | Evaluated at 24 months in both arms compared to enrollment (baseline) data
  75% reduction in seizure frequency
Seizure freedom in response to first prescribed anti-epileptic drug | 6 months after enrollment of final subject
  Percentage of children seizure free for 6 months or longer in response to the first anti-epileptic drug prescribed, as measured by questions in standardized case report forms completed by physicians with epilepsy expertise, blinded as to the arm of the study. The blinded physicians will review a daily seizure log which indicates the occurrence and duration of each seizure, maintained by the parent/guardian, to facilitate the blinded physician evaluation.
Diagnostic accuracy | Evaluated by blinded physicians at 1, 6, 12, 18, and 24 months after enrollment
  Diagnostic accuracy among study subjects in both arms, determined by blinded physicians
Mortality | Once, at study conclusion (24 months after enrollment of final subject)
  Differences in mortality between study arms that cannot be explained by potential differences in disease severity
Status epilepticus | Assessed at 1 month, 6 months, 12 months, 18 months and 24 months after enrollment, with analysis of outcome at study conclusion (24 months after enrollment of final subject)
  Difference in frequency of episodes of status epilepticus among children in both arms of the study, as measured by questions in standardized case report forms completed by physicians with expertise in epilepsy, who are blinded as to the arm of the study. The blinded physicians will review a daily seizure log which indicates estimated seizure duration for each seizure, maintained by the parent/guardian, to facilitate the blinded physician evaluation.
Morbidity | Once, at study conclusion (24 months after enrollment of final subject)
  Differences in morbidity, including neurodevelopmental morbidity, associated with epilepsy between study arms that emerged during the cRCT
Diagnostic tests ordered | Once, at study conclusion (24 months after enrollment of final subject)
  Differences by study arm in number and type of diagnostic tests (e.g., MRIs, EEGs) ordered
Task-shifted protocol adherence | Once, at study conclusion (24 months after enrollment of final subject)
  Percentage adherence by CHWs to protocol in the task-shifted arm
Anytime 6-month seizure-free interval | Assessed at 4 time points during 24-month follow-up: 6, 12, 18, and 24 months
  6-month seizure-free intervals as determined by evaluations by physicians with expertise in epilepsy, blinded as to the arm of the study, at 6 months, 12 months, 18 months and 24 months after enrollment. These blinded physicians with expertise in epilepsy will record seizure frequency (including seizure-freedom) on standardized case report forms, facilitated by blinded physician review of daily seizure logs maintained by parents/guardians that will indicate the specific dates and durations of all recorded seizures.

OTHER OUTCOMES:
Cost-effectiveness of task-shifted care | Data collection over 24 months after enrollment, with analysis of cost-effectiveness data after the final study subject completes the 24-month follow-up visit.
  Comparison of total financial epilepsy care costs between task-shifted and enhanced usual care study arms, as measured at specified intervals throughout both arms of the study - 1 week, 1 month, 2 months, 4 months, 6 months, 9 months, 12 months, 18 months, and 24 months after enrollment through questions about care received in standardized case report forms, and with financial costs determined by health economists who verify costs of care at specific private and government healthcare facilities.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Trevathan, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Aminu Taura, MBBS, Principal Investigator — Aminu Kano Teaching Hospital
Locations (3):
- Nigeria (3):
  - Federal Neuro-Psychiatric Hospital, Kaduna
  - Aminu Kano Teaching Hospital, Kano
  - Ahmadu Bello University Teaching Hospital, Zaria

IPD SHARING:
Plan to Share IPD: Yes
The principal investigators and research personnel will share deidentified data from the study in multiple modes:
  1. Data files for internal (study) investigators
  2. Data files for external (non-study) investigators
  3. Timely and comprehensive publication of the results for the primary and secondary outcomes
  4. Public-access data files supplied to NIH
Supporting Information: Study Protocol
Time Frame: A standard analysis file will be created for use in the analysis of the trial, and for manuscripts and reports. At the end of the trial, the analysis file will be circulated to each internal investigator. If an internal trial investigator requests a special file be created for him/her, a complete proposal must be submitted as detailed below. The contents/variables of the standard analysis file will be posted in the members-only section of the trial website. The internal analysis file will include data from screening and baseline forms, follow-up visit forms with CHWs, seizure diaries, medication administration diaries, neurological exams, laboratory (clinical laboratory, EEG, brain imaging) forms, and outcomes. A section for potential external investigators will also be created on the trial website, which will list the variables from the case report forms. In general, external investigators will be limited to variables from this list.
Access Criteria: Both internal and external investigators are required to submit a proposal requesting a dataset from the trial, describing the following elements in detail:
  1. Investigator's name and affiliation
  2. Hypothesis to be tested or investigation to be conducted
  3. Background and relevant literature
  4. Subjects eligible for inclusion in the analysis and dataset
  5. List of variables of interest
  6. Substantially detailed analysis plan
  7. List of potential co-authors and collaborators

REFERENCES:
- [Background] de Boer HM, Moshe SL, Korey SR, Purpura DP. ILAE/IBE/WHO Global Campaign Against Epilepsy: a partnership that works. Curr Opin Neurol. 2013 Apr;26(2):219-25. doi: 10.1097/WCO.0b013e32835f2037. PMID 23449175
- [Background] de Boer HM, Mula M, Sander JW. The global burden and stigma of epilepsy. Epilepsy Behav. 2008 May;12(4):540-6. doi: 10.1016/j.yebeh.2007.12.019. Epub 2008 Feb 14. PMID 18280210
- [Background] Diop AG, de Boer HM, Mandlhate C, Prilipko L, Meinardi H. The global campaign against epilepsy in Africa. Acta Trop. 2003 Jun;87(1):149-59. doi: 10.1016/s0001-706x(03)00038-x. PMID 12781390
- [Background] Ndoye NF, Sow AD, Diop AG, Sessouma B, Sene-Diouf F, Boissy L, Wone I, Toure K, Ndiaye M, Ndiaye P, de Boer H, Engel J, Mandlhate C, Meinardi H, Prilipko L, Sander JW. Prevalence of epilepsy its treatment gap and knowledge, attitude and practice of its population in sub-urban Senegal an ILAE/IBE/WHO study. Seizure. 2005 Mar;14(2):106-11. doi: 10.1016/j.seizure.2004.11.003. PMID 15694563
- [Background] Mbuba CK, Ngugi AK, Fegan G, Ibinda F, Muchohi SN, Nyundo C, Odhiambo R, Edwards T, Odermatt P, Carter JA, Newton CR. Risk factors associated with the epilepsy treatment gap in Kilifi, Kenya: a cross-sectional study. Lancet Neurol. 2012 Aug;11(8):688-96. doi: 10.1016/S1474-4422(12)70155-2. Epub 2012 Jul 6. PMID 22770914
- [Background] Newton CR, Garcia HH. Epilepsy in poor regions of the world. Lancet. 2012 Sep 29;380(9848):1193-201. doi: 10.1016/S0140-6736(12)61381-6. PMID 23021288
- [Background] Wilmshurst JM, Cross JH, Newton C, Kakooza AM, Wammanda RD, Mallewa M, Samia P, Venter A, Hirtz D, Chugani H. Children with epilepsy in Africa: recommendations from the International Child Neurology Association/African Child Neurology Association Workshop. J Child Neurol. 2013 May;28(5):633-44. doi: 10.1177/0883073813482974. Epub 2013 Mar 28. PMID 23539548
- [Background] Wilmshurst JM, Kakooza-Mwesige A, Newton CR. The challenges of managing children with epilepsy in Africa. Semin Pediatr Neurol. 2014 Mar;21(1):36-41. doi: 10.1016/j.spen.2014.01.005. Epub 2014 Jan 14. PMID 24655403
- [Background] Mbuba CK, Newton CR. Packages of care for epilepsy in low- and middle-income countries. PLoS Med. 2009 Oct;6(10):e1000162. doi: 10.1371/journal.pmed.1000162. Epub 2009 Oct 13. PMID 19823570
- [Background] Mbuba CK, Ngugi AK, Newton CR, Carter JA. The epilepsy treatment gap in developing countries: a systematic review of the magnitude, causes, and intervention strategies. Epilepsia. 2008 Sep;49(9):1491-503. doi: 10.1111/j.1528-1167.2008.01693.x. Epub 2008 Jun 13. PMID 18557778